CLINICAL TRIAL: NCT01247727
Title: Clinical Application of Multimodal Physiological Signal Analysis in Critical Ill Patients Depending on Extracorporeal Membrane Oxygenation
Brief Title: Heart Rate Variability in Extracorporeal Membrane Oxygenation (ECMO) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Je Ko/National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 201010075R
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Heart Rate Variability
Keywords: Heart rate variability; extracorporeal membrane oxygenation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
National Taiwan University Hospital is the leading center for care of patients with extracorporeal membrane oxygenation (ECMO). The predictable factors associated with outcomes are still lacking in patients with the ECMO support. The aim of this study is to collect the electrical signals stored in the monitor of intensive care units (ICUs), which are analyzed by the bio-informatics software. The pre-, peri-, and post-ECMO heart rate variability, including linear and non-linear analysis is calculated to address the association with outcomes of patients with ECMO. In addition, we collected the demographics, body temperature, respiratory rate, and blood pressure to investigate the causes of heart rate variability.

DETAILED DESCRIPTION:
Inclusion criteria:Adults patients (aged older than 18 years; less than 90 years old) used ECMO for cardiopulmonary support

Exclusion criteria:

1. Patients used illicit drugs
2. Patients received heart transplantation
3. Patients have the history of arrhythmia

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (aged > 18 years; less than 90 years old) used ECMO for cardiopulmonary support

Exclusion Criteria:

* Patients used illicit drugs
* Patients received heart transplantation
* Patients have the history of arrhythmia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with the support of extracorporeal membrane oxygenation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Je Ko, M.D., Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan